CLINICAL TRIAL: NCT05846152
Title: Study of the Concordance of the Measurements Between the Evaluation of the Area of a Wound by the Technique of Transparent (Gold Standard) Compared to the Evaluation of the Area by the Algorithm of a Decision Support System (Wound-size)
Acronym: PIXAIRE_I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, MAXANT Guillaume, Principal investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-A01546-37
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Wound Healing
Keywords: Wound; Healing; Surface; Tissue content
MeSH Terms: conditions — Wounds and Injuries | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WoundCare medical device (Experimental): Unique arm. The patients undergo all interventions planned in the study.
  Interventions: Device: Intervention

INTERVENTIONS:
Device: Intervention — Patient wounds will be examined:
  * by eye by the principal investigator
  * using a ruler by the principal investigator
  * by WoundCare algorithms (AKA WoundTrack) using smartphone photography by the principal investigator
  * by eye by a second investigator
  * using a ruler by a second investigator
  * by WoundCare (AKA WoundTrack) algorithms using smartphone photography by a second investigator.

SUMMARY:
The goal of this clinical trial is to compare the evaluation of a wound area and wound tissue content made by different methods on patient population with need for directed wound healing.

The main question test of the concordance of the measurements between the evaluation of the area of a wound by the technique of transparent (Gold standard) compared to the evaluation of the area by the algorithm of a decision support system (WoundSize)

Patient wounds will be examined:

* by eye by the principal investigator
* using a ruler by the principal investigator
* by WoundCare algorithms (AKA WoundTrack) using smartphone photography by the principal investigator
* tracing the outline of the wound using a transparent sheet by the principal investigator
* by eye by a second investigator
* using a ruler by a second investigator
* by WoundCare (AKA WoundTrack) algorithms using smartphone photography by a second investigator.
* tracing the outline of the wound using a transparent sheet by the second investigator

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a wound requiring controlled healing ranging from 4 to 150 cm²
* Age greater than or equal to 18 years old
* Person affiliated to a social security scheme or beneficiary of such a scheme
* Person having received complete information on the organization of the research and having signed informed consent.
* Wound that can be taken in one photo in its entirety.

Exclusion Criteria:

* Person with a medical condition which, in the judgment of the investigator, is not compatible with participation in the study
* Wound on a part of the body that would make the person participating in the photos of the wound identifiable (tattoo, piercing, birthmark, etc.).
* Several wounds are in the photo.
* Pregnant, parturient or breastfeeding women
* Person deprived of liberty by a judicial or administrative decision
* Adult subject to a measure of legal protection (guardianship, curatorship, safeguard of justice) or unable to express their consent, persons subject to psychiatric care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-05-02 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
WoundCare (AKA WoundTrack) the principal investigator | During the study inclusion visit
  Surface (cm2) is evaluated using the software WoundCare (AKA WoundTrack) the principal investigator
Transparent sheet by principal investigator | During the study inclusion visit
  Surface (cm2) is evaluated tracing the outline of the wound using a transparent sheet by the principal investigator

SECONDARY OUTCOMES:
Eye by the principal investigator | During the study inclusion visit
  Surface (cm2) is evaluated by the eye of the principal investigator
Ruler by the principal investigator | During the study inclusion visit
  Surface (cm2) is evaluated using a ruler by the principal investigator
Eye by the second investigator | During the study inclusion visit
  Surface (cm2) is evaluated by the eye of the second investigator
Ruler by the second investigator | During the study inclusion visit
  Surface (cm2) is evaluated using a ruler by the second investigator
WoundCare (AKA WoundTrack) the second investigator | During the study inclusion visit
  Surface (cm2) is evaluated using the software WoundCare (AKA WoundTrack) the second investigator
Transparent sheet by second investigator | During the study inclusion visit
  Surface (cm2) is evaluated tracing the outline of the wound using a transparent sheet by the second investigator

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Maxant, Dr, Principal Investigator — HAGUENAU Hospital

IPD SHARING:
Plan to Share IPD: No